CLINICAL TRIAL: NCT02672826
Title: Description of the Endothelial Phenotypes From the Subcutaneous Abdominal and Gluteo-femoral Adipose Tissues in Women
Acronym: ADIPENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12 067 08
Record Dates: First submitted 2016-01-11; First posted 2016-02-03 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adipose tissue surgery (Experimental): The adipose tissue surgery (gluteo-femoral and abdominal) will be obtained from women programmed for surgery in which the estrogenic status as well as adipose tissue mass profile will be evaluated.
  Interventions: Procedure: Adipose tissue surgery

INTERVENTIONS:
Procedure: Adipose tissue surgery — Adipose tissue (gluteo-femoral and abdominal) will be obtained from women programmed for surgery in which the estrogenic status as well as adipose tissue mass profile will be evaluated

SUMMARY:
The endothelium is a key barrier between blood and tissue compartments. It is a major target of factors involved in metabolic and cardiovascular pathologies. However, the study of native human adult endothelial cells is difficult due to the lack of appropriate models and thereafter the endothelium is actually not easily accessible for clinical investigation. However, our results recently showed that the endothelium from human adipose tissue exhibit distinct phenotypes, including endothelial cell number and inflammatory, angiogenic and senescent state, according to adipose tissue location, i.e. subcutaneous and visceral. It is well recognized that estrogens favour gluteo-femoral adipose tissue deposit and their deficit after menopause is associated with increased abdominal and visceral fat mass as well as metabolic dysfunctions. These perturbations might be prevented with hormonal therapy. However, no data are available concerning the endothelial cells from gluteo-femoral and abdominal adipose tissues in women.

DETAILED DESCRIPTION:
The adipose tissues (gluteo-femoral and abdominal) will be obtained from women programmed for surgery in which the estrogenic status as well as adipose tissue mass profile will be evaluated. The phenotype (inflammatory and angiogenic activation and senescent state) of native endothelial cells will be determined "in situ" by immunohistochemical and flow cytometry approaches and on isolated endothelial cells by Reverse transcriptase-Q Polymerase Chain Reaction and Western blot. In vitro approaches will be performed 1) to establish a causal relationship between endothelial senescence and activation state, 2) to define the impact of the adipose tissue microenvironment on the endothelial cell activation and senescence and 3) to study the potential protective effect of estrogens on endothelial senescence.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight for at least 3 months
* Women undergoing a surgery of subcutaneous adipose tissue

Exclusion Criteria:

* Undergoing Insulin therapy
* Undergoing steroidal and nonsteroidal anti-inflammatory treatments
* undergoing or stopped since less than 6 months immunosuppressive treatments
* Positive serology for HIV, Hepatitis B Virus and/or Hepatitis C Virus

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-04-24 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
number of endothelial cells | day 1

SECONDARY OUTCOMES:
number of senescent cells | day 1
Correlation between estrogens level on endothelial senescence | day 1
Correlation between endothelial senescence and activation state | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois ARNAL, MD PhD, Principal Investigator — Explorations Fonctionnelles physiologiques
Locations (1):
- Explorations fonctionnelles Physiologiques - Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aupetit A, Decaunes P, Belles C, Riant E, Galitzky J, Chapouly C, Laisne M, Flores-Flores R, Chaput B, Vie K, Arnal JF, Bouloumie A, Briot A. Endothelial DLL4 Is an Adipose Depot-Specific Fasting Sensor Regulating Fatty Acid Fluxes. Arterioscler Thromb Vasc Biol. 2023 May;43(5):684-696. doi: 10.1161/ATVBAHA.122.318876. Epub 2023 Mar 16. PMID 36924232